CLINICAL TRIAL: NCT05740020
Title: Effect of Virtual Reality in Spider Cage on Gross Motor Performance and Balance in Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amr Mohsen Mohamed Abo Khatwa (Other)
Responsible Party: Sponsor-Investigator, Amr Mohsen Mohamed Abo Khatwa, bachelor's degree of physical therapy, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EG, KFS lab Research 1
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): Group (A) will receive virtual reality in addition to the traditional exercise program.
  Interventions: Device: virtual reality glasses; Other: The traditional exercise program
- Group (B) (Active Comparator): Group (B) will receive traditional exercise program.
  Interventions: Other: The traditional exercise program

INTERVENTIONS:
Device: virtual reality glasses — A specialized VR glasses will be used and VR games application in spider cage
  Arms: Group (A)
Other: The traditional exercise program — The selected physical therapy program:
  1. Neurodevelopmental approach: aims to facilitate typical motor development and function and to prevent secondary impairments (figure 4).
  2. Approximation: aims to control spasticity and stimulate the joint mechanoreceptors (figure 5).
  3. Stretching exercise: aims to maintain length and flexibility of shorten muscles (figure 6).
  4. Strengthening exercise: aims to improve the functional ability (figure 7).
  5. Spider suspension exercise for 30 minutes (figure 8).
  5. Gait training activities: aims to improve balance (figure 9). 6. Balance training program: aims to improve balance (figure 10).

SUMMARY:
This study will detect the effect of virtual reality in spider cage on gross motor performance and balance in children with spastic diplegia.

DETAILED DESCRIPTION:
The current study will be directed to investigate effect of virtual reality on gross motor and balance as the weakness of the trunk muscles and lower limb muscles along with spasticity potentially predispose balance and walking issues of children with bilateral spastic CP .

The balance deficits in children with CP are multifactorial. According to the system's model proposed by Woollacott and Shumway-Cook, multiple systems contribute to postural dysfunction in children with CP. Muscle weakness and stiffness of lower limb muscles account for biomechanical constraints and postural malalignment during standing and functional balancing.

Virtual reality is one of the novel technology-based approaches to treat balance and motor function in children with CP. It utilizes the interactive simulations created in computer hardware and software, in which the children find opportunities to engage in environments appearing real to them .

After reviewing the available previous published studies, it was found that there is no previous study directly compared between the effects of virtual reality and physical therapy in spider cage on gross motor performance and balance with diplegic children CP children. Both therapeutic modalities were found to induce good clinical outcomes when studied separately, so this study will be conducted to examine the effectiveness of virtual reality.

The greater demand for physical therapy for Paediatrics' signifies the need for more effective, safer and evident therapeutic modalities. The findings of this study will help both; the therapists and the children to save time, effort and reach the best results in concise times.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included in the study if they fulfil the following criteria:

  1. A medical diagnosis of spastic diplegic CP made by pediatricians or pediatric neurologists.
  2. Children with spasticity grades ranged from 1 to 2+ according to Modified Ashworth scale (MAS).
  3. Their age range from 6 to 12 years.
  4. Children who can sit on the chair with good balance and recognize and follow verbal orders and commands included in both testing and training techniques.

Exclusion Criteria:

* Children with a permanent spastic diplegia, who might have one or more of the following, will be excluded:

  1. They had a permanent deformity (bony or soft tissue contractures).
  2. Children having visual or auditory defects.
  3. Current hospitalization for urgent medical reasons.
  4. Severe mental retardation.
  5. Children who will undergo fewer than twelve regular sessions of physical therapy at their place will not be included in the survey.
  6. Children with history of epileptic seizure or any diagnosed cardiac or orthopedic disability that may hinder assessment methods and treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
GROSS MOTOR PERFORMANCE | 3 monthes
  we will use Gross Motor Function Measure 88 (GMFM-88) to measure Gross motor performance.
  this score range from (0 to 100 ) zero is the minimum value and 100 is the maximum value
BALANCE | 3 monthes
  we will use Pediatric Balance Scale (PBS) to measure Balance. this score range from (0 to 56 ) zero is the minimum value and 56 is the maximum value

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT05740020/Prot_SAP_ICF_000.pdf